CLINICAL TRIAL: NCT02824445
Title: A Pilot Study to Evaluate the Efficacy of EEG/ECG-guided Magnetic Resonant Therapy (MeRT) in War Veterans With Posttraumatic Stress Disorder (PTSD) at Tinker and MacDill Air Force Bases
Brief Title: To Evaluate the Efficacy of EEG-guided Magnetic Resonant Therapy in War Veterans With Posttraumatic Stress Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to permanant change of stations of investigators.
Sponsor: 72nd Medical Group, Tinker Air Force Base (U.S. Federal Agency)
Collaborators: brain treatment center; MacDill AFB (Unknown)
Responsible Party: Principal Investigator, Jianzhong Zhang, Chief, Aeromedical Services, 72nd Medical Group, Tinker Air Force Base
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FWH20150038H
Record Dates: First submitted 2016-06-23; First posted 2016-07-06 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Post-Traumatic Stress Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham (Sham Comparator): The double-blind is used during the first 2 weeks. From week 3 and on, the study becomes open label. Subjects in Group I (active MeRT treatment group) will continue receive active MeRT treatment for W3/4; subjects in Group II (placebo/sham group) will receive active MeRT treatment from W3 to W6 for 4 weeks. All subjects will receive 4 weeks active MeRT treatment. The study ends in 8th wk. The data collection points are baseline, weeks of 2, 4, 6, and 8. The data from weeks 1-2 (Phase I) will be utilized to analyze the safety and any effect of MRT procedure may have over placebo. The data from weeks 3 on (Phase II) will be used to address if any benefit of longer MeRT treatment (4 vs 2 weeks). The study design offers both groups 4 weeks of the experimental therapy in a row. This will provide potentially equal benefit to those participants assuming that MeRT helps to improve PTSD symptoms.
  Interventions: Device: individualized Transcranial Magnetic Stimulation
- Treatment (Experimental): The double-blind is used during the first 2 weeks. From week 3 and on, the study becomes open label. Subjects in Group I (active MeRT treatment group) will continue receive active MeRT treatment for W3/4; subjects in Group II (placebo/sham group) will receive active MeRT treatment from W3 to W6 for 4 weeks. All subjects will receive 4 weeks active MeRT treatment. The study ends in 8th wk. The data collection points are baseline, weeks of 2, 4, 6, and 8. The data from weeks 1-2 (Phase I) will be utilized to analyze the safety and any effect of MRT procedure may have over placebo. The data from weeks 3 on (Phase II) will be used to address if any benefit of longer MeRT treatment (4 vs 2 weeks). The study design offers both groups 4 weeks of the experimental therapy in a row. This will provide potentially equal benefit to those participants assuming that MeRT helps to improve PTSD symptoms.
  Interventions: Device: individualized Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: individualized Transcranial Magnetic Stimulation
  Other Names: EEG-GUIDED MAGNETIC RESONANT THERAPY (MeRT)

SUMMARY:
After 13 years of war, PTSD has become pervasive in service members. Traditionally it is evaluated by PTSD Checklist Military Version (PCL-M) and treated with cognitive processing therapy, prolonged exposure therapy and medication management with limited success. Repetitive Transcranial Magnetic Stimulation (TMS) has shown efficacy for improving individual cognitive function in the past decades, both in healthy population and in patients with depression. TMS has been approved by the FDA in treatment of major depressive disorder and migraine headaches. Magnetic EEG guided Resonant Treatment (MeRT) is a form of individualized TMS based on member's EEG/ECG input. Investigators propose to use MeRT to treat veterans with war-related PTSD, a syndrome that includes depressive and anxious symptoms; it is likely that MeRT (namely TMS) will be beneficial and comparable to or better than the current FDA approved methods for treating PTSD.

ELIGIBILITY:
Inclusion Criteria:

1. Have diagnosis of combat-related PTSD by DSM-V criteria, diagnosed via clinical interview by psychologist or psychiatrist (note: combat pilots of remotely piloted aircraft are included)
2. PCL-M score > 45
3. Age between 18 and 55 years (at day of informed consent)
4. Willing and able to adhere to the treatment schedule and all required study visits.
5. Must be clinically stable for at least 30 days on or off any PTSD medication before the trial treatment

Exclusion Criteria:

1. Individuals diagnosed by the Investigator with the following conditions (current unless otherwise stated):

   * History of open skull traumatic brain injury
   * History of clinically significant seizure disorder
2. Individuals with a clinically defined neurological disorder including, but not limited to:

   * Any condition likely to be associated with increased intracranial pressure
   * Space occupying brain lesion
   * History of cerebrovascular accident
   * Cerebral aneurysm
3. Abnormalities that indicate risk of seizure, i.e., focal or general slowing or spikes during EEG recording
4. Any type of rTMS treatment within 3 months prior to the screening visit
5. Currently under antipsychotic medication treatment
6. Intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, stents, or electrodes) or any other metal object within or near the head, excluding the mouth, which cannot be safely removed
7. Clinically significant abnormality or clinically significant unstable medical condition that in the Investigator's judgment might pose a potential safety risk to the subject or limit interpretation of the trial results
8. Clinically significant medical illness, including any uncontrolled thyroid disorders, hepatic, cardiac, pulmonary and renal malfunctioning
9. Any condition which in the judgment of the investigator would prevent the subject from completion of the study
10. Inability to acquire a clinically satisfactory EEG/ECG on a routine basis
11. Grossly abnormal electrolyte or cell blood count panels suggestive of other pathology at study initiation
12. Pregnant or breastfeeding women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2018-05-28 (Actual)

PRIMARY OUTCOMES:
The outcome will be measured by PTSD checklist -- military version (PCL-M) scoring criteria for PTSD. The outcome is measured additionally by Cognitive and Physical Functioning Questionnaire (CPFQ) for cognitive function improvement among the subjects. | At the end of week of 4 and 8.
  The change of PCL-M and CPFQ scores from baseline and at weeks of 4 and 8 are assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- 72d Medical Group, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes